CLINICAL TRIAL: NCT01617928
Title: A Phase 1 Study of Veliparib (ABT-888) in Combination With Carboplatin/Paclitaxel in Japanese Subjects With Solid Tumors
Brief Title: A Study of Veliparib in Combination With Carboplatin and Paclitaxel in Japanese Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-629
Record Dates: First submitted 2012-05-23; First posted 2012-06-13 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2013-07

CONDITIONS: Solid Tumors
MeSH Terms: interventions — veliparib; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- veliparib (ABT-888) (Experimental)
  Interventions: Drug: veliparib (ABT-888); Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: veliparib (ABT-888) — Dosing orally twice daily starting Day 1 through day 7 of each cycle. Decisions to move to the next cohort will be based on evaluation of DLTs in the current cohort. Decisions will be made with a discussion between the Sponsor and the principal investigator to dose escalate or de-escalate or add more subjects to the cohort.
Drug: carboplatin — Carboplatin will be administered on Day 3 of each cycle, intravenously.
  Other Names: paraplatin
Drug: paclitaxel — Paclitaxel will be administered on Day 3 of each cycle, intravenously.
  Other Names: taxol

SUMMARY:
This is a Phase 1 open-label study and consists of 3 treatment groups (dose levels) . Treatment cycles are 3 weeks in duration. The primary objective of this study is to determine the recommended phase two dose (RPTD) of veliparib (ABT-888) when administered in combination with carboplatin and paclitaxel in Japanese subjects with solid tumors. Secondary objectives are to assess pharmacokinetics and to obtain a preliminary efficacy of anti-tumor activity in the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed malignant solid tumor.
* Patients who are amenable to standard combination chemotherapy of carboplatin and paclitaxel.
* Patients should have received less than or equal to 1 prior chemotherapy regimens for advanced stage disease.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Patients must have normal organ and marrow function

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or the adverse events due to agents administered more than 3 weeks earlier have not recovered to less than grade 2.
* Known history of allergic reactions to carboplatin or cremophor-paclitaxel.
* Patients who have previously received a poly(ADP-ribose) polymerase (PARP) inhibitor.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active systemic infection requiring treatment, symptomatic congestive heart failure, angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of seizure disorder.
* Hepatitis B surface antigen (HBsAg) positive, Hepatitis C virus (HCV) antibody positive or Human immunodeficiency virus (HIV)-positive patients.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose and recommended Phase two dose | During the first cycle (21 days from first dose of veliparib)

SECONDARY OUTCOMES:
Pharmacokinetics; Area Under the Curve (AUC), Maximum observed plasma concentration (Cmax) and Time to Cmax (Tmax) of veliparib (ABT-888) | Eight timepoints on Day 1 of first cycle (21 days)
Pharmacokinetics; Area Under the Curve (AUC), Maximum observed plasma concentration (Cmax) and Time to Cmax (Tmax) of veliparib (ABT-888) when administered in combination with carboplatin and paclitaxel | Eight timepoints on Day 3 of first cycle (21 days)
Pharmacokinetics; Area Under the Curve (AUC), Maximum observed plasma concentration (Cmax) and Time to Cmax (Tmax) of paclitaxel when administered in combination with veliparib (ABT-888) and carboplatin | Eight timepoints on Day 3 of first cycle (21 days)
Pharmacokinetics; Area Under the Curve (AUC), Maximum observed plasma concentration (Cmax) and Time to Cmax (Tmax) of carboplatin when administered in combination with veliparib (ABT-888) and paclitaxel | Six timepoints on Day 3 of first cycle (21 days)
Preliminary tumor response | From date of first dose of veliparib until the date of first documented progression or date of death from any cause, whichever come first, assessed up to 6 cycles.
  Computerized tomography (CT) scan of chest, abdomen and pelvis to assess tumor burden
Safety assessment; Physical exam including vital signs | From date of first dose of veliparib until 30 days after last dose of veliparib (up to 6 cycles)
  Blood pressure, pulse and body temperature
Safety assessment; Clinical lab testings | From date of first dose of veliparib until 30 days after last dose of veliparib (up to 6 cycles)
  Hematology, Chemistry and Urinalysis
Safety assessment; Adverse event monitoring | From date of first dose of veliparib until 30 days after last dose of veliparib (up to 6 cycles)
  Collect all adverse events at each visit
Safety assessment; Change from Baseline in Electrocardiogram (ECG) | Day 8 of first cycle (21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Hideyuki Hashiba, BS, Study Director — AbbVie
Locations (1):
- Site Reference ID/Investigator# 68622, Tokyo, Japan

REFERENCES:
- [Result] Mizugaki H, Yamamoto N, Nokihara H, Fujiwara Y, Horinouchi H, Kanda S, Kitazono S, Yagishita S, Xiong H, Qian J, Hashiba H, Shepherd SP, Giranda V, Tamura T. A phase 1 study evaluating the pharmacokinetics and preliminary efficacy of veliparib (ABT-888) in combination with carboplatin/paclitaxel in Japanese subjects with non-small cell lung cancer (NSCLC). Cancer Chemother Pharmacol. 2015 Nov;76(5):1063-72. doi: 10.1007/s00280-015-2876-7. Epub 2015 Oct 3. PMID 26433581